CLINICAL TRIAL: NCT01941654
Title: A Single-arm Phase II Study to Determine the Efficacy of Preemptive Local Ablative Therapy to Residual Metabolic Active Oligo-metastases in Those EGFR Mutation Positive Non-small Cell Lung Cancer Patients Who Have Achieved a Good Partial Response With First-line EGFR TKI (ATOM)
Brief Title: ATOM_local Ablative Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Cancer Trials Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN060
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: NSCLC; Activating EGFR Mutation

STUDY DESIGN:
Intervention Model Description: RT + Oral TKI
Oversight: Data Monitoring Committee: No

ARMS (1):
- preemptive local ablative therapy (Experimental)
  Interventions: Radiation: preemptive local ablative therapy; Drug: Oral TKI

INTERVENTIONS:
Radiation: preemptive local ablative therapy
Drug: Oral TKI

SUMMARY:
To determine the efficacy of preemptive local ablative therapy in NSCLC patients with activating EGFR mutation who have oligometastatic residual metabolic-active disease after first-line EGFR TKI, as measured by PFS rate at 1 year from the trial enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed UICC 7th edition Stage IIIB (not amenable for curative intent local radiotherapy)/IV (metastatic or recurrent) non-small cell carcinoma of lung
2. Documented activating EGFR mutation (exon 19 deletion or exon 21 L858R only) in tumor tissues
3. Treated with first-line EGFR TKI for 3 months and achieved good radiological partial response that was documented with a CT scan
4. Not more than 4 residual metabolic active (SUVmax > 2.5) metastatic sites left on the screening PET-CT scan. (one bone metastatic site is regarded as a single site, mediastinal/ hilar lymph nodes in close proximity and possible to be treated in an acceptable volume is regarded as one lesion)
5. The shortest diameter of the lesion must be ≥ 1cm and is amenable to local ablative therapy
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
7. Age ≥ 18 years
8. Pleural or pericardial effusion at diagnosis is allowed only if it has resolved on CT scan after 3-month EGFR TKI treatment
9. Brain metastasis at diagnosis is allowed if it has been treated either surgically or with radiotherapy and there is no radiological progression on follow-up CT scan. The patient is neurologically stable for at least 1 week after cessation of steroid treatment
10. Adequate organ function as defined by the following criteria:

    1. Serum alanine transaminase ≤ 3 x upper limit of normal (ULN) or ≤ 5 x ULN if liver function abnormalities are due to liver metastases
    2. Total bilirubin ≤ 1.5 x ULN
    3. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    4. Platelets count ≥ 100 x 109/L
    5. Creatinine clearance > 45ml/min
11. Written informed consent that is consistent with ICH-GCP guidelines

Exclusion Criteria:

1. Prior chemotherapy is not allowed except adjuvant chemotherapy for completely resected early staged non-small cell lung cancer and it has been at least 12 months before the start of EGFR TKI treatment
2. Prior radiotherapy is not allowed except brain irradiation
3. Leptomeningeal carcinomatosis
4. Lymphangitis carcinomatosis of lung
5. Prior or concomitant malignancy at other sites is not allowed except treated non-metastatic non-melanoma skin cancer, ductal carcinoma-in-situ of breast and carcinoma-in-situ of cervix with curative intent
6. Uncontrolled active infection or medical condition (e.g. uncontrolled hypertension, unstable angina, congestive heart failure [≥ NYHA Class II], uncontrolled arrhythmia, myocardial infarction or cerebrovascular accident within the past 6 month)
7. Pre-existing interstitial lung disease
8. Woman of child-bearing potential or male patient is unwilling to use adequate birth control method prior to the study entry, for the duration of study participation and for at least 2 months after the EGFR TKI treatment has ended.
9. Pregnant and Lactating female patient
10. Non-compliance to the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09-18 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
PFS rate at 1 year | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Progression-free survival | 2 years
radiologic change on PET-CT scan 3 months after SABR | 3 months
Number of Participants with Adverse Events as a Measure of safety | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kwok Chi LAM, FRCP, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Department of Clinical Oncology, Hong Kong, Hong Kong